CLINICAL TRIAL: NCT07167563
Title: Real-world Lithium Intake Measured by a Pillbox: A Clinical Study to Test Real-world Compliance With Lithium Treatment
Brief Title: Real-world Lithium Intake
Status: Recruiting | Type: Observational
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Other Study IDs: 2025_01_eLi12
Record Dates: First submitted 2025-08-29; First posted 2025-09-11 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-08

CONDITIONS: Bipolar Disorder (BD)
Keywords: Lithium
MeSH Terms: conditions — Bipolar Disorder | interventions — Lithium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with bipolar disorder treated with lithium
  Interventions: Other: Lithium (LI) based on clinical indication

INTERVENTIONS:
Other: Lithium (LI) based on clinical indication — Participants have for 4 weeks a pill box registering the time for lithium intake. Weekly phone calls will assess whether patients can remember the time for lithium intake.

SUMMARY:
The aim of the present study is to study compliance with lithium therapy and patterns of lithium intake among a representative group of patients with bipolar disorder in a real-world clinical setting. This will be studied via a pill box that registers the daily time when the participant took the lithium tablet out of the pill box, representing a proxy for the actual lithium intake. Participants will receive a weekly phone call asking for several aspects of lithium intake.

DETAILED DESCRIPTION:
Bipolar disorder is a severe mental disorder1 and lithium represents the first-line pharmacological treatment1-5. The individual lithium dose is based on monitoring of clinical effect and lithium blood levels6,7 (i.e., plasma lithium (P-Li) levels), which can be measured easily and accurately via blood sampling. Treatment guidelines recommend measuring P-Li levels during up-titration, but also regularly (2-4x/year) when patients have reached a stable dose6-8. P-Li levels are also measured to avoid high blood levels that are associated with side effects. Specifically, it is well-known that lithium can have adverse effects on the kidneys9-11 and the thyroid gland11, and that the therapeutic window is relatively narrow6.

P-Li levels reach a peak concentration after 2-4 hours, following which the concentration steadily decreases, as lithium is excreted entirely through the kidneys6. Treatment guidelines have for >50 years recommended that P-Li levels should be measured 12 hours after the patient has taken the most recent lithium dose in order to evaluate the target P-Li and lithium dose for each individual patient6,7,12, allowing a time window from 10 to 14 hours after lithium intake6,7,13,14. Typically, patients take the lithium dose in the evening and the blood sample is collected the following morning before a potential morning dose of lithium is taken. As the vast majority of lithium-treated patients are outpatients, this 12-hour timing depends entirely on the patient, meaning that the patient is responsible to get the blood test 12 hours after the most recent lithium intake. However, patients may have difficulties to get the lithium blood test taken 12 hours after the lithium dose15, blood sampling may be delayed for logistic reasons, and/or patients forget about the specific timing. Hence, P-Li levels may not necessarily reflect the actual 12-hour P-Li level and this complicates clinical decision-making. Indeed, initial data from Central Denmark Region have indicated that 50-75% of lithium-treated patients may not comply with the 12-hour lithium blood test requirement16. This has a potential high impact as e.g., a P-Li level measured 16 hours after the last lithium dose, but interpreted as a 12-hour P-Li level, may lead to an unwarranted increase of the lithium dose, potentially increasing the risk for side effects.

We have developed a new method to estimate the 12-hour P-Li level, termed eLi12 (estimated lithium level at 12 hours). eLi12 is a mathematical equation that can estimate the 12-hour P-Li when the lithium blood test is taken at a different time point, e.g., 8 or 16 hours. This method would represent a solution for the abovementioned clinical challenge but depends on the patient-reported time for lithium intake. As the time point of the lithium blood test always is registered, eLi12 depends on that the patient takes the prescribed lithium dose and correctly reports the time for intake of the most recent lithium intake before the lithium blood test. However, despite that the self-reported time for lithium intake has been used for >50 years in everyday clinical treatment, no study has investigated the pattern on lithium intake in a real-world clinical setting.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years
2. Diagnosed with bipolar disorder (ICD-10: F30-31)
3. Followed at the bipolar disorder outpatient clinic at AUHP
4. Treated with lithium (ATC-code: N05AN01)
5. Able to give informed oral and written consent.

Exclusion Criteria:

1. Any coercive measure in the study period including patients in forensic psychiatry.
2. In a clinical condition where the treating clinician evaluates that the patient is not able to attend the research study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any patient aged ≥18 years diagnosed with bipolar disorder followed at the bipolar disorder outpatient unit at AUHP, treated with lithium and without any coercive measure or forensic psychiatry sanction at the time of inclusion will be eligible for inclusion in the study.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-07-05 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-07-15 (Estimated)

PRIMARY OUTCOMES:
Compliance with lithium therapy | From enrollment for 4 weeks
  Study if patients take their lithium medication on a daily basis, which is measured via a pillbox that registers the time for lithium intake (used for 4 weeks by each participant)
Regular intake | From enrollment for 4 weeks
  Study whether lithium-treated patients take their lithium medication at the same time of day, meaning within 30 minutes of the same time point (measured for 4 weeks via a pillbox containing the lithium medication)
The mean time in minutes between the self-reported time for intake of the most recent lithium dose (mentioned at the weekly phone call) and the registered time for the actual intake of the most recent lithium dose (i.e., the most recent intake of lithium | From enrollment for 4 weeks
If a larger deviation between the self-reported and the registered time for lithium intake (i.e. the measure from co-primary outcome 3) depends on if participants are in a (hypo)manic or depressive mood state (which is answered at the weekly phone call). | From enrollment for 4 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Clinic for Bipolar Disorder, Aarhus University Hospital Psychiatry, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No
Not possible due to local data protection rules.